CLINICAL TRIAL: NCT03020147
Title: Follow-up of Low Birth Weight Cohort of 2008-2013
Brief Title: Low Birth Weight Follow-up
Status: Completed | Type: Observational
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Other Study IDs: BandimHP
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Non Specific Effects of Vaccine; Bacillus-Calmette-Guerin; Low Birth Weight; Maternal Immunisation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- early BCG: Children received BCG soon after their birth between 2008 and 2013.
- delayed BCG: Children received BCG when they are 2,5kg between 2008 and 2013.

SUMMARY:
The Randomized Control Trail included 4,172 low-birth weight children between February 2008 and September 2013 in Bissau. The children who were included in the RCT and who are living in the Bandim Health Project study area will be visited. The study assistants will ask about the health of the child and of both parents. Furthermore, Bacille Calmette-Guerin (BCG) scar status of both child and parents will be checked.

ELIGIBILITY:
Inclusion Criteria:

* Participation during the low birth weight BCG trial between 2008 and 2013.

Exclusion Criteria:

* Not living in the Bandim Health Project's study area.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children who participated in the low birth weight trial between 2008 and 2013.
Sampling Method: Probability Sample
Enrollment: 1258 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
mortality differences between group who received early BCG and late BCG | up to 8 years of age
mortality by parental scar status | up to 8 years of age

SECONDARY OUTCOMES:
hospitalization rate between early BCG and late BCG group | last two weeks
consultation rate between early BCG and late BCG group | last two weeks
medication use between early BCG and late BCG group | last two weeks

OTHER OUTCOMES:
hospitalization based on parental scar status | last two weeks
consultations based on parental scar status | last two weeks
medication use based on parental scar status | last two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Bissau, Bissau Codex, Guinea-Bissau

REFERENCES:
- [Background] Aaby P, Roth A, Ravn H, Napirna BM, Rodrigues A, Lisse IM, Stensballe L, Diness BR, Lausch KR, Lund N, Biering-Sorensen S, Whittle H, Benn CS. Randomized trial of BCG vaccination at birth to low-birth-weight children: beneficial nonspecific effects in the neonatal period? J Infect Dis. 2011 Jul 15;204(2):245-52. doi: 10.1093/infdis/jir240. PMID 21673035
- [Background] Biering-Sorensen S, Aaby P, Napirna BM, Roth A, Ravn H, Rodrigues A, Whittle H, Benn CS. Small randomized trial among low-birth-weight children receiving bacillus Calmette-Guerin vaccination at first health center contact. Pediatr Infect Dis J. 2012 Mar;31(3):306-8. doi: 10.1097/INF.0b013e3182458289. PMID 22189537